CLINICAL TRIAL: NCT07265596
Title: Early Longitudinal Imaging in the Parkinson's Progression Markers Initiative Using [18F] AV-133 (PPMI AV-133 Prodromal Imaging)
Brief Title: Early Longitudinal Imaging in the Parkinson's Progressive Marker Initiative (PPMI) Using (18F)AV-133 (PPMI AV-133 Prodromal Imaging)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PPMI 015
Record Dates: First submitted 2025-09-12; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Prodromal Parkinsons Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Prodromal Parkinson's disease (PD) (Experimental): Prodromal Parkinson's disease participants enrolled in the PPMI Clinical 002 study will receive 3 injections of [18F] AV-133 and imaging procedures over the course of 24 months.
  Interventions: Drug: [18F] AV-133 PET Imaging

INTERVENTIONS:
Drug: [18F] AV-133 PET Imaging — Prodromal PD participants from the PPMI Clinical (002) study will be followed for up to 24 months. These participants will undergo imaging assessments with [18F]AV-133 under this protocol at baseline, 12-month and 24 months.

SUMMARY:
The study is a longitudinal, multi-center study to assess progression of [18F] AV-133 imaging in Prodromal PD participants. Participants will be followed for up to 24 months. Approximately 100 Prodromal participants will be recruited from up to 10 sites. Participants will be comprehensively assessed at baseline and follow up. Participants will undergo imaging assessments with [18F] AV-133 and clinical (motor, neuropsychiatric, cognitive and imaging and biomarker) assessments (conducted under the PPMI Clinical protocol).

DETAILED DESCRIPTION:
The Parkinson's Progression Marker Initiative (PPMI) is an observational, international, multi-center study designed to identify PD progression biomarkers both to improve understanding of disease etiology and course and to provide the necessary tools to enhance the likelihood of success of therapeutics studies to slow PD progression (ClinicalTrials.gov Identifier: NCT01141023). A key focus of PPMI is to identify biomarkers during the period when PD neurodegeneration is already present, but symptoms of PD have not yet occurred. This prodromal cohort would enable us to investigate PD biomarker signatures prior to onset of typical symptoms of PD. The study is a longitudinal, multi-center study to assess progression of [18F]AV-133 imaging in Prodromal PD participants. The PPMI 015 study will enroll participants from the PPMI Clinical (002) study. Participants will be followed annually for up to 24 months.

Approximately 100 Prodromal participants will be recruited from up to 10 sites. Participants will be comprehensively assessed at baseline and follow up.

Participants will undergo [18F]AV-133 PET imaging targeting the vesicular monoamine transporter. All participants will undergo an initial [18F]AV-133 PET imaging scan at baseline with repeat imaging at 12 months and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. A Prodromal PD participant, over the age of 18, confirmed as eligible to proceed to PPMI Clinical Baseline visit.
2. Able to provide informed consent.
3. Male or Female (females must meet additional criteria specified below as applicable)

   * Females must be of non-childbearing potential or using a highly effective method of birth control 14 days prior to until at least 24 hours after injection of 18F-AV-133

     * Non-childbearing potential is defined as a female that must be either postmenopausal (no menses for at least 12 months prior to PET scan) or surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy).
     * Highly effective method of birth control is defined as practicing at least one of the following: A birth control method that results in a less than 1% per year failure rate when used consistently and correctly, such as oral contraceptives for at least 3 months prior to injection, an intrauterine device (IUD) for at least 2 months prior to injection, or barrier methods, e.g., diaphragm or combination condom and spermicide. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) is not acceptable.
   * Females of childbearing potential must not be pregnant, breastfeeding or lactating.

     * Includes a negative urine pregnancy test prior to injection of 18F-AV-133 on day of PET scan.

Exclusion Criteria:

1. Received any of the following medications that might interfere with 18F- AV-133 PET imaging: tetrabenazine (TBZ) or methylphenidate, reserpine, or amphetamine derivative, within 1 month prior to the Baseline 18F-AV-133 injection.
2. Any other medical or psychiatric condition or lab abnormality, which in the opinion of the investigator might preclude participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
[18F]AV-133 mean rate of change and variability | 24 months
  The mean rates of change and the variability around the mean of [18F]AV-133 PET SUVr in Prodromal PD patients, and where appropriate the comparison of these rates between patient subsets at study intervals ranging from 12 months to 24 months.

SECONDARY OUTCOMES:
[18F]AV-133 prediction of clinical motor progression | 24 months
  Predictive value of [18F]AV-133 imaging Standardized Uptake Value ratio [SUVr] at baseline for longitudinal clinical progression, defined as change in Movement Disorder Society sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS), scale [0-260]
[18F]AV-133 prediction of clinical cognitive progression | 24 months
  Predictive value of [18F]AV-133 imaging Standardized Uptake Value ratio [SUVr] at baseline for longitudinal cognitive progression, defined as change in cognitive scales Montreal Cognitive Assessment (MoCA), scale [0-30]
[18F]AV133 cutoff for clinical PD | 24 months
  Determine [18F]AV-133 SUVr cutoff value for predicting development of clinical diagnosis of PD in people with Prodromal PD.
  Compare [18F]AV-133 SUVr with DaTscan SBR cutoffs for predicting the development of clinical diagnosis of PD in people with Prodromal PD.
[18F] AV133 correlation with DaTscan | 24 months
  Correlation between the longitudinal change of [18F]AV-133 and DaTscan.
Correlation of [18F]AV133 change with change in clinical and biomarker outcomes | 24 months
  Correlation between the longitudinal change of imaging outcomes and MDS-UPDRS, other clinical and blood biomarkers and sensor outcomes.
Incidence of Treatment emergent adverse events | 24 months
  Number of participants with treatment-related adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Ken Marek, MD, Principal Investigator — Institute for Neurodegenerative Disorders
Locations (8):
- United States (2):
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - University of Pennsylvania, Philadelphia, Pennsylvania
- Toronto Western Hospital, Toronto, Ontario, Canada
- Philipps-University of Marburg, Hessen, Germany
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Radboud University, Nijmegen, Gelderland, Netherlands
- United Kingdom (2):
  - Queen Mary University of London, London, Britain
  - Newcastle University, Newcastle upon Tyne, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Undecided